CLINICAL TRIAL: NCT00062660
Title: An Open Label Safety Study to Evaluate the Safety of Tipranavir Plus Ritonavir When Used in Combination With Other Agents for the Treatment of Patients With HIV Infection Who Have Failed and/or Are Intolerant to Combination Antiretroviral Therapy and Have Limited Treatment Options
Brief Title: Tipranavir in Patients With Progressive, Systemic HIV-1 Disease Who Have Failed or Are Intolerant to Currently Approved Treatments for HIV Infection
Status: Approved for marketing | Type: Expanded Access
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1182.58
Record Dates: First submitted 2003-06-10; First posted 2003-06-12 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir

INTERVENTIONS:
Drug: Tipranavir — Tipranavir 250 mg soft elastic capsules

SUMMARY:
To provide early access to tipranavir and evaluate the safety and tolerance of tipranavir combined with low dose of ritonavir in patients with progressive, HIV-1 disease who have failed or are intolerant to currently approved treatments for HIV infection, who are unable to participate in another tipranavir controlled clinical trial and have an urgent need for anti-HIV treatment.

ELIGIBILITY:
Inclusion criteria:

Patients aho have a positive serology HIV antibody test confirmed by Western blot, p24 antigen assay, HIV-1 RNA or HIV culture and are highly pre-treated and virus resistant to multiple protease inhibitors.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (146):
- United States (35):
  - 1182.58.31, Scottsdale, Arizona
  - 1182.58.29, Los Angeles, California
  - 1182.58.34 Campus Code 696446, Los Angeles, California
  - 1182.58.42 Synergy Hematology/Oncology, Los Angeles, California
  - 1182.58.43, Los Angeles, California
  - 1182.58.03, San Francisco, California
  - 1182.58.33 Kaiser Permanente Medical Center, Clinical Trials Unit, San Francisco, California
  - 1182.58.37 AIDS Health Care Foundation, Los Angeles, Connecticut
  - 1182.58.41 Circle Medical, LLC, Norwalk, Connecticut
  - 1182.58.28, Washington D.C., District of Columbia
  - 1182.58.38, Miami Beach, Florida
  - 1182.58.40 Drs. Raben and Feldman Research Associates, South Miami, Florida
  - 1182.58.23 Hillsborough County Health Department, Tampa, Florida
  - 1182.58.36 Suite 525, Atlanta, Georgia
  - 1182.58.08, Honolulu, Hawaii
  - 1182.58.22, Chicago, Illinois
  - 1182.58.32, New Orleans, Louisiana
  - 1182.58.15, Boston, Massachusetts
  - 1182.58.19 Henry Ford Hospital, Detroit, Michigan
  - 1182.58.04 Kansas City Free Health Clinic, Kansas City, Missouri
  - 1182.58.25 Wohl Clinic, St Louis, Missouri
  - 1182.58.02 Wellness Center, Las Vegas, Nevada
  - 1182.58.09 Polari Medical Group, New York, New York
  - 1182.58.30, Chapel Hill, North Carolina
  - 1182.58.06 University of Cincinnati Medical Center, Infectious diseases, Cincinnati, Ohio
  - 1182.58.35, Portland, Oregon
  - 1182.58.14, Philadelphia, Pennsylvania
  - 1182.58.20 University of Pittsburgh, Pittsburgh, Pennsylvania
  - 1182.58.01 Boehringer Ingelheim Investigational Site, Columbia, South Carolina
  - 1182.58.10 Comprehensive Care Center, Nashville, Tennessee
  - 1182.58.18 University of Texas Southwest Medical Center at Dallas, Dallas, Texas
  - 1182.58.07, Houston, Texas
  - 1182.58.039 Olmos Park Medical Associates, San Antonio, Texas
  - 1182.58.11 Swedish Medical Center, Seattle, Washington
  - 1182.58.44 VW Hospital and Clinics, Madison, Wisconsin
- Australia (25):
  - 1182.58.61005 Royal Prince Alfred Hospital, Camperdown, New South Wales
  - 1182.58.61008 St Vincents Hospital, Darlinghurst, New South Wales
  - 1182.58.61011 St Vincents Hospital, Darlinghurst, New South Wales
  - 1182.58.61014 St Vincents Hospital, Darlinghurst, New South Wales
  - 1182.58.61007 407 Doctors Pty Ltd, Darlinghusrst, New South Wales
  - 1182.58.61019 407 Bouke Street, Darlinghusrst, New South Wales
  - 1182.58.61022 Sexual Health Clinic, Kingswood, New South Wales
  - 1182.58.61012 Bigge Park Centre, Liverpool, New South Wales
  - 1182.58.61003 The Prince of Wales Hospital, Randwick, New South Wales
  - 1182.58.61002 Royal North Shore Hospital, St Leonards, New South Wales
  - 1182.58.61006 Albion Street Clinic, Surry Hills, New South Wales
  - 1182.58.61025 Immunology Department, Westmead, New South Wales
  - 1182.58.61010 Biala Building, Brisbane, Queensland
  - 1182.58.61009 Level 6, Herston, Queensland
  - 1182.58.61024, Nambour, Queensland
  - 1182.58.61016 Princess Alexandra Hospital, Woolloongabba, Queensland
  - 1182.58.61020, Adelaide, South Australia
  - 1182.58.61015 Flinders Medical Centre, Bedford Park, South Australia
  - 1182.58.61001 88 Rathdowne Street Carlton, Carlton, Victoria
  - 1182.58.61018 Melbourne Sexual Health Clinic, Carlton, Victoria
  - 1182.58.61017 Department of Infectious Diseases, Clayton, Victoria
  - 1182.58.61013 Melbourne Sexual Health Clinic, Melbourne, Victoria
  - 1182.58.61023, Melbourne, Victoria
  - 1182.58.61021, South Yarra, Victoria
  - 1182.58.61004 Royal Perth Hospital, Perth, Western Australia
- Belgium (4):
  - 1182.58.3201 Boehringer Ingelheim Investigational Site, Antwerp
  - 1182.58.3202 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.58.3203 Boehringer Ingelheim Investigational Site, Brussels
  - 1182.58.3204 Boehringer Ingelheim Investigational Site, Liège
- Denmark (3):
  - 1182.58.4505 Aarhus Universitetshospital Skejby, Aarhus C
  - 1182.58.4501 Rigshospitalet, København Ø
  - 1182.58.4504 Odense Universitetshospital, Odense C
- France (34):
  - 1182.58.33029 Hôpital Aix, Aix-en-Provence
  - 1182.58.33001 Hôpital Saint Jacques, Besançon
  - 1182.58.33022 Hôpital Avicenne, Bobigny
  - 1182.58.33020 Hôpital Antoine Beclère, Clamart
  - 1182.58.33028 Hôpital Louis Mourier, Colombes
  - 1182.58.33027 Hôpital, Dijon
  - 1182.58.33034 Hôpital Raymond Poincarré, Garches
  - 1182.58.33006 Hôpital Bicêtre, Le Kremlin-Bicêtre
  - 1182.58.33019 Hôpital de l'Hôtel Dieu, Lyon
  - 1182.58.33031 Hôpital edouard Herriot, Lyon
  - 1182.58.33009 Hôpital de la Conception, Marseille
  - 1182.58.33023 Hôpital Sainte Marguerite, Marseille
  - 1182.58.33030 Hôpital Saint Eloi, Montpellier
  - 1182.58.33032 Hôpital Emile Muller, Mulhouse
  - 1182.58.33008 Hôpital Hôtel Dieu, Nantes
  - 1182.58.33003 Hôpital de l'Archet, Nice
  - 1182.58.33005 Hôpital Bichat, Paris
  - 1182.58.33007 Hôpital Georges Pompidou, Paris
  - 1182.58.33013 Hôpital Saint Louis, Paris
  - 1182.58.33014 Hôpital Cochin, Paris
  - 1182.58.33017 Hôpital Bichat Claude Bernard, Paris
  - 1182.58.33018 Hôpital Saint Antoine, Paris
  - 1182.58.33024 Hôpital Necker, Paris
  - 1182.58.33033 Hôpital Tenon, Paris
  - 1182.58.33035 Hôpital des Abîmes, Pointe à Pitre
  - 1182.58.33012 Hôpital Robert Debré, Reims
  - 1182.58.33026 Hôpital Ponchaillou, Rennes
  - 1182.58.33015 Hôpital Civil, Strasbourg
  - 1182.58.33025 Hôpital Foch, Suresnes
  - 1182.58.33021 Hôpital Chalucet, Toulon
  - 1182.58.33002 Hôpital Purpan, Toulouse
  - 1182.58.33016, Tourcoing
  - 1182.58.33010 Hôpital Brabois, Vandœuvre-lès-Nancy
  - 1182.58.33011 Hôpital Paul Brousse, Villejuif
- 1182.58.3001, Athens, Greece
- Ireland (2):
  - 1182.58.44016 St James Hospital, Dept of Genito Urinary Medicine, Dublin
  - 1182.58.44029 Our Lady For Sick Children, Dublin
- Italy (8):
  - 1182.58.3903 Università di Brescia, Brescia
  - 1182.58.3904 Ospedali Riuniti di Foggia, Foggia
  - 1182.58.3901 Ospedale Luigi Sacco, Milan
  - 1182.58.3902 Ospedale L. Sacco, Milan
  - 1182.58.3907 Presidio Ospedaliero di Rimini, Rimini
  - 1182.58.3905 Presidio Dalmati, S. Angelo Lodigiano (lo)
  - 1182.58.3906 Ospedale Infantile Regina Margherita, Torino
  - 1182.58.3908 Centro Medicina Preventiva, Verona
- 1182.58.35102 Hospital Condes Castro Guimarães, Cascais, Portugal
- South Africa (5):
  - 1182.58.27095 Boehringer Ingelheim Investigational Site, Cape Town
  - 1182.58.27098 Boehringer Ingelheim Investigational Site, Cape Town
  - 1182.58.27099 Boehringer Ingelheim Investigational Site, Cape Town
  - 1182.58.27096 Boehringer Ingelheim Investigational Site, Durban
  - 1182.58.27097 Boehringer Ingelheim Investigational Site, Westville, Durban
- Switzerland (6):
  - 1182.58.4101 Boehringer Ingelheim Investigational Site, Basel
  - 1182.58.4103 Boehringer Ingelheim Investigational Site, Bern
  - 1182.58.4104 Boehringer Ingelheim Investigational Site, Geneva
  - 1182.58.4107 Boehringer Ingelheim Investigational Site, Geneva
  - 1182.58.4102 Boehringer Ingelheim Investigational Site, Zurich
  - 1182.58.4105 Boehringer Ingelheim Investigational Site, Zurich
- United Kingdom (22):
  - 1182.58.44020 Beckenham Hospital, Beckenham
  - 1182.58.44004 Boehringer Ingelheim Investigational Site, Brighton
  - 1182.58.44002 Boehringer Ingelheim Investigational Site, Cardiff
  - 1182.58.44025 Boehringer Ingelheim Investigational Site, Chertsey
  - 1182.58.44019 Boehringer Ingelheim Investigational Site, Chichester
  - 1182.58.44009 Boehringer Ingelheim Investigational Site, Edinburgh
  - 1182.58.44023 Boehringer Ingelheim Investigational Site, Harrow
  - 1182.58.44024 Boehringer Ingelheim Investigational Site, Leeds
  - 1182.58.44003 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44005 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44008 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44010 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44014 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44017 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44018 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44026 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44027 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44028 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44031 Boehringer Ingelheim Investigational Site, London
  - 1182.58.44011 Boehringer Ingelheim Investigational Site, Peterborough
  - 1182.58.44022 Boehringer Ingelheim Investigational Site, Woolwich
  - 1182.58.44030 Boehringer Ingelheim Investigational Site, Woolwich